CLINICAL TRIAL: NCT05322369
Title: Prevalence of Periodontitis in Diabetic Patients of Egyptian Population : A Cross Sectional Study.
Brief Title: Prevalence of Periodontitis in Diabetic Patients of Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Reda Refaiy Basuony, Prevalence of periodontitis in diabetic patients of Egyptian population : A cross sectional study., Cairo University
Other Study IDs: Periodontitis in diabetics
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Periodontitis; Diabetes
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: periodontal charting only — Periodontal charting only

SUMMARY:
The study aims at determining the prevalence of Periodontitis in diabetic Egyptian dental outpatients attending the diagnostic centre at faculty of Dentistry, Cairo University

DETAILED DESCRIPTION:
Periodontitis is a common chronic inflammatory disease which is characterized by destruction of the supporting structures of the teeth especially the periodontal ligament and alveolar bone. Their classification is complex and takes into consideration many factors such as the clinical presentation, age at diagnosis, rate of disease progression, and systemic and local factors which may increase risk (Pihlstrom BL etal., 2005).

Tissue destruction in periodontitis results in the breakdown of the collagen fibers of the periodontal ligament, that results in the formation of a periodontal pocket between the gingiva and the tooth. "Pocketing" is not evident on simple visual inspection, and assessment using a periodontal probe is needed. Periodontitis is a slowly progressing disease, however the tissue destruction that happens is largely irreversible. The condition is asymptomatic in the early stages, it is not usually painful, and many patients are unaware till progression in the condition occurs and is enough to result in tooth mobility. As a result of the further destruction of fibers of the periodontal ligament (referred to as attachment loss), the pockets deepen, and the resorption of the alveolar bone occurs in parallel with the progressing attachment loss (Grossi SG etal., 1995).

Diabetes mellitus is a metabolic disorder which is characterized by hyperglycemia as a result of defective secretion or activity of insulin (Tan M etal., 1997). It may be further complicated by poor regulation of protein and lipid metabolism. In the current classification of this condition, the terms "insulin-dependent diabetes mellitus" and "non-insulin dependent diabetes mellitus" are not used, in part because they relate to treatment rather than to the diagnosis. A conclusive diagnosis of diabetes mellitus is done through assessment of glycated hemoglobin levels. In those people with diabetes, sequential fasting plasma glucose levels will be 7 mmol/L or more.

Type 1 diabetes mellitus normally occurs as a result of destruction of the beta cells in the islets of Langerhans of the pancreas by the autoimmune system. This condition often leads to absolute deficiency of insulin. Type 1 diabetes tends to occur in young, lean individuals, usually before 30 years of age; however, older patients may also present with this form of diabetes occasionaly.

With Type 2 diabetes, patients can still produce insulin but do so relatively inadequately. In many cases, the pancreas produces larger than normal quantities of insulin. A major feature of Type 2 diabetes is a lack of sensitivity to insulin by the cells of the body, especially fat and muscle cells. These larger quantities of insulin are produced as an attempt to get these cells to recognize that insulin is present.

There is emerging evidence to support the existence of a two-way relationship between diabetes and periodontitis, with diabetes increasing the risk for periodontitis, and periodontal inflammation negatively affecting glycemic control (Fox CH., 1992) & (Mealey BL & Ocampo GL, 2007).

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients whether Type 1 or 2
* Patient consulting in the outpatient clinic
* Provide informed consent.

Exclusion Criteria:

* Participants who had <10 teeth currently or
* Those who had undergone any periodontal treatment within the past 1 year
* Patients suffering from any other metabolic or systemic diseses tht could affect the periodontal condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic Egyptian patients attending the outpatient diagnostic center of the faculty of dentistry, Cairo University
Sampling Method: Non-Probability Sample
Enrollment: 447 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-03-02 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
: Prevalence of Periodontitis in diabetics of Egyptian outpatients of faculty of dentistry cairo university. | Baseline
  periodontal charting will be done for diabetic patients attending outpatient clinics

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud R Reda, BDS, Principal Investigator — Cairo University
Locations (1):
- Faculty of dentistry cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided